CLINICAL TRIAL: NCT00742690
Title: Terlipressin Given As I.V. Boluses Vs Terlipressin Given As Continuous Intravenous Infusion In Patients With Cirrhosis And Type 1 Hepatorenal Syndrome (Hrs): Preliminary Results Of A Randomized Controlled Clinical Study.
Brief Title: Terlipressin Given As I.V. Boluses Versus Terlipressin Given As Continuous Intravenous Infusion In Patients With Cirrhosis And Type 1 Hepatorenal Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Responsible Party: Clinica Medica 5, Univeristy of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1442P
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Cirrhosis; Type 1 Hepatorenal Syndrome
Keywords: cirrhosis; type 1 hepatorenal syndrome; terlipressin; albumin; effective circulating volume; Patients; with
MeSH Terms: conditions — Fibrosis | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 35 patients with cirrhosis and type 1 HRS
  Interventions: Drug: terlipressin given by intravenous boluses and albumin
- 2 (Experimental): 35 patients with cirrhosis and type 1 HRS
  Interventions: Drug: terlipressin given by continuous intravenous infusion and albumin

INTERVENTIONS:
Drug: terlipressin given by intravenous boluses and albumin — Patients who will be randomly assigned to arm 1 will received terlipressin given by intravenous boluses at the initial dose of terlipressin was 0.5 mg/4 hr. In case of non response, the dose of terlipressin was progressively increased up to a maximum of 2 mg/4 hr. Human albumin will be given intravenously at the dose of 1 g/kg of body weight on the first day followed by 20-40 g/day.
  Arms: 1
Drug: terlipressin given by continuous intravenous infusion and albumin — Patients who will be randomly assigned to arm 1 will received terlipressin given as intravenous boluses at the initial dose of 0.5 mg/4 hr. In case of non response, the dose of terlipressin will be progressively increased up to a maximum of 2 mg/4 hr. Human albumin will be given at the dose of 1 g/kg of body weight at the first day followed by 20-40 g/day.
  Arms: 2

SUMMARY:
It is well known that terlipressin and albumin improve renal function in patients with cirrhosis and type 1 HRS. In previous studies terlipressin has been used either as intravenous boluses moving from an initial dose of 0.5-1 mg/4 hr or as continuous intravenous infusion at the initial dose of 2 mg/24 h. Up to now the two schedules of i.v. administration of terlipressin have never been compared. Nevertheless, it has been hypothesized that continuous intravenous infusion assures a more steady profile of effect on portal pressure in patients with cirrhosis. Thus, the aim of the study will be to compare terlipressin given as i.v. bolus vs terlipressin given as continuous intravenous infusion in the treatment of type 1 HRS in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis and type 1 HRS

Exclusion Criteria:

* HCC beyond the Milan Criteria,septic shock (systolic arterial pressure < 90 mmHg,
* Significant heart or respiratory failure,
* Peripheral arteriophaty clinically significant,
* Previous heart stroke or significant alteration of the ECG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-05; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
The primary end-point of the study is the complete reform of the renal function (creatinine < 1.5 mg/dl). | The treatment will be continued for a maximum of 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Unit, General Hospital, Padua, Italy

REFERENCES:
- [Result] Angeli P, Guarda S, Fasolato S, Miola E, Craighero R, Piccolo F, Antona C, Brollo L, Franchin M, Cillo U, Merkel C, Gatta A. Switch therapy with ciprofloxacin vs. intravenous ceftazidime in the treatment of spontaneous bacterial peritonitis in patients with cirrhosis: similar efficacy at lower cost. Aliment Pharmacol Ther. 2006 Jan 1;23(1):75-84. doi: 10.1111/j.1365-2036.2006.02706.x. PMID 16393283